CLINICAL TRIAL: NCT02080598
Title: Cigarette and Gastric Contents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lionel Bouvet (Other)
Responsible Party: Sponsor-Investigator, Lionel Bouvet, Doctor, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Allocation: Randomized | Model: Crossover
Other Study IDs: 2014-A00127-40; L14-12 (Other: Comité de Protection des Personnes Sud Est IV)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Variation of the Antral Area After Cigarettes Smoking or Not

ARMS (2):
- Controle (No Intervention): The volunteer do not smoke any cigarette during the study period
- smoking (Experimental): the volunteer smokes 2 cigarettes in 15 minutes
  Interventions: Behavioral: 2 cigarettes in 15 minutes

INTERVENTIONS:
Behavioral: 2 cigarettes in 15 minutes
  Arms: smoking

SUMMARY:
The aims of this cross over prospective study are to demonstrate that smoking two cigarettes do not change the gastric contents and volume in fasting volunteers.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 Volunteers habitual smokers = 5 cigarettes / day during at least 1 year

Exclusion Criteria:

* Digestive Diseases, gastroparesis
* Non smokers
* pregnancy
* history of diabetes mellitus
* medication affecting gastric motility
* previous gastrointestinal surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Variation of the ultrasonographically measured antral area afer smoking or non smoking cigarette | every 30 minutes during 2h30

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Lazaar S, Boselli E, Chassard D, Allaouchiche B, Bouvet L. Effect of acute cigarette smoking on gastric contents in regular smoker volunteers. A prospective randomized cross-over study. Br J Anaesth. 2015 Oct;115(4):590-4. doi: 10.1093/bja/aev264. Epub 2015 Aug 30. PMID 26323291